CLINICAL TRIAL: NCT01561352
Title: An Open Label Pilot Study to Test the Efficacy and Safety of Recombinant Factor VIIa (rFVIIa, NovoSeven®) in the Treatment of Refractory Hemorrhagic Cystitis Following High Dose Chemotherapy
Brief Title: Efficacy and Safety of Activated Recombinant Human Factor VII in Refractory Haemorrhagic Cystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F7HAEM-2080
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Other Haemostasis Disorder; Haemorrhagic Cystitis
MeSH Terms: conditions — Cystitis, Hemorrhagic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Factor VII (Experimental)
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII — If non-responding haemorrhagic cystitis to 24-hour trial of conventional therapy, 80 mcg/kg is administered i.v. for the first dose. If necessary, two additional doses of 120 mcg/kg can be administered i.v.

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to assess the efficacy of activated recombinant human factor VII in the treatment of refractory haemorrhagic cystitis (HC) following chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Severe haemorrhagic cystitis (HC)

Exclusion Criteria:

* Patients with overt DIC (disseminated intravascular coagulation)
* Patients with known active atherosclerotic disease, such as active coronary artery disease or recent stroke in the past 3 months
* Central venous access device related thrombus in the last 3 months
* Patients with allergy to activated recombinant human factor VII or any component of its preparation

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2001-09; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Reduction of hematuria that failed 24-hour standard therapy evaluated by change of urine color
Reduction of hematuria that failed 24-hour standard therapy evaluated by urine haemoglobin content
Reduction of hematuria that failed 24-hour standard therapy evaluated by urocrit

SECONDARY OUTCOMES:
Symptoms of venous or arterial thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Houston, Texas

REFERENCES:
- [Result] Ashrani AA, Gabriel DA, Gajewski JL, Jacobs DR Jr, Weisdorf DJ, Key NS. Pilot study to test the efficacy and safety of activated recombinant factor VII (NovoSeven) in the treatment of refractory hemorrhagic cystitis following high-dose chemotherapy. Bone Marrow Transplant. 2006 Dec;38(12):825-8. doi: 10.1038/sj.bmt.1705535. No abstract available. PMID 17133240
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com